CLINICAL TRIAL: NCT01540773
Title: Growth Hormone 120 Minutes Following a Single Low-dose of Amino Acids in Healthy Subjects.
Brief Title: Single Low-Dose of Supplement Amino Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PBRC 10043
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Growth Hormone; Amino Acid
Keywords: growth hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- amino acid supplement (Active Comparator): supplements with the proprietary amino acid derivative blend.
  Interventions: Drug: Amino acid supplement
- Placebo (Placebo Comparator): Non-Active
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amino acid supplement — An orally administered supplement of the proprietary amino acid derivative
  Other Names: SeroVital™
  Arms: amino acid supplement
Drug: Placebo — A non-active orally administered supplement of the proprietary amino acid derivative
  Other Names: non-active
  Arms: Placebo

SUMMARY:
The purpose of the study is to confirm the results of a prior study that demonstrated pills containing two amino acids which are in foods increased growth hormone and insulin-like growth factor-1.

DETAILED DESCRIPTION:
Oral supplementation with a key combination of derivatives that has been shown to increase human growth hormone in healthy volunteers peaking at 90 minutes and IGF-1 at 8 hours post-administration.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and healthy females
* Between 18 and 70 years

Exclusion Criteria:

* Pregnant or nursing
* Taking any chronic medication including birth control pills.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Tam CS, Johnson WD, Rood J, Heaton AL, Greenway FL. Increased Human Growth Hormone After Oral Consumption of an Amino Acid Supplement: Results of a Randomized, Placebo-Controlled, Double-Blind, Crossover Study in Healthy Subjects. Am J Ther. 2020 Jul/Aug;27(4):e333-e337. doi: 10.1097/MJT.0000000000000893. PMID 30893070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were Volunteers at Pennington Biomedical Research Center, Baton Rouge, LA USA, between October 2011 and March 2011.
Pre-assignment Details: 16 participants recruited; 16 Screened, 0 excluded
Groups:
- Amino Acid Supplement, Then Placebo: 50% of participants first received an orally administered supplement with the proprietary amino acid derivative blend. After a washout period of one week, they then received a Placebo tablet (matching the amino acid supplement).
- Placebo, Then Amino Acid Supplement: 50% of participants first received an orally administered Placebo tablet (matching the amino acid supplement). After a washout period of one week, they then received the orally administered supplement with the proprietary amino acid derivative blend.
Period: First Intervention
Arm/Group | Amino Acid Supplement, Then Placebo | Placebo, Then Amino Acid Supplement
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Wash Out Period of 1 Week
Arm/Group | Amino Acid Supplement, Then Placebo | Placebo, Then Amino Acid Supplement
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Amino Acid Supplement, Then Placebo | Placebo, Then Amino Acid Supplement
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Crossover of amino acid supplement to placebo or placebo to amino acid supplement
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Growth Hormone
Description: Measure human growth hormone at times 0-120 minutes on two occasions about one week apart. On one occasion, the proprietary amino acid derivative blend will be given orally at time 0 in capsule form, and on the other occasion the capsules will contain no amino acids.
Time Frame: 0-120 minutes, at Baseline and post dose, week 1 and week 3
Measure: Mean (95% Confidence Interval); unit: nanograms/ml
Groups:
- Amino Acid Supplement: supplements with the proprietary amino acid derivative blend.
  Amino acid supplement: An orally administered supplement of the proprietary amino acid derivative
  A single dose of amino acids can significantly increase GH levels after 120 minutes in healthy men and women. Whether these GH changes persist over a longer duration or have other positive effects is being further examined.
Arm/Group | Amino Acid Supplement | Placebo
Number analyzed (Participants) | 16 | 16
nanograms/ml | 1.15 [0.17 to 2.14] | -0.48 [-1.47 to 0.50]
Statistical Analysis 1: Comparison: Amino Acid Supplement vs Placebo; Test type: Superiority; p = 0.01, t-test, 2 sided

2. Primary Outcome: Area Under the Curve of Growth Hormone Over Baseline
Description: as for outcome 1
Time Frame: 0-120 minutes, at Baseline and post dose, week 1 and week 3
Measure: Mean (95% Confidence Interval); unit: min*ng/mL
Groups:
- Amino Acid Supplement: Participants received an orally administered supplement with the proprietary amino acid derivative blend.
- Placebo: Participants received an orally administered Placebo tablet (matching the amino acid supplement).
Arm/Group | Amino Acid Supplement | Placebo
Number analyzed (Participants) | 16 | 16
min*ng/mL | 20.43 [19.9 to 20.95] | 19.67 [18.74 to 20.59]
Statistical Analysis 1: Comparison: Amino Acid Supplement vs Placebo; Test type: Superiority; p = 0.04, t-test, 2 sided

3. Secondary Outcome: Insulin-like Growth Factor 1
Description: Measure IGF-1 8 hours following the administration of the capsules containing the proprietary amino acid derivative blend or placebo
Time Frame: 8 hours following administration
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Amino Acid Supplement | Placebo
Number analyzed (Participants) | 16 | 16
ng/mL | 208.125 (55.769) | 224.375 (67.903)

ADVERSE EVENTS:
Arm/Group | Amino Acid Supplement | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amino Acid Supplement (N=16) | Placebo (N=16)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No